CLINICAL TRIAL: NCT00955292
Title: A Phase I, Multicenter, Open-label, Dose-Escalation, Safety, Pharmacokinetic and Pharmacodynamic Study of Quarfloxin Administered Intravenously Weekly for Three Weeks of a Four Week Cycle in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: Dose-escalation Study of Quarfloxin in Patients With Advanced Solid Tumors or Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Modified dose schedule presented no advantage over previously studied schedule
Sponsor: Cylene Pharmaceuticals (Industry)
Responsible Party: C. Padgett, Cylene Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3-07-002
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Advanced Solid Tumors; Lymphoma
Keywords: Solid Tumors; Lymphoma; G-Quadruplex
MeSH Terms: conditions — Lymphoma | interventions — CX 3543

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quarfloxin (Experimental)
  Interventions: Drug: Quarfloxin

INTERVENTIONS:
Drug: Quarfloxin — Escalating doses of quarfloxin administered intravenously for 24 hours once weekly for three weeks every four weeks
  Other Names: CX-3543; Quarfloxacin

SUMMARY:
This phase 1 study of quarfloxin (CX-3543) is designed to test the safety, tolerability, and highest safe dose of this drug when administered intravenously weekly for three weeks of a four week cycle in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Quarfloxin is a first-in-class small-molecule targeted cancer therapeutic derived from the validated fluoroquinolone class of drugs. Quarfloxin was rationally designed to target a G-quadruplex (QPLX) DNA structure and disrupt protein-DNA interactions essential to cancer cells. The QPLX targeted by quarfloxin forms within ribosomal DNA (rDNA) and the QPLX is bound by the nucleolin protein.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed solid tumors or lymphomas.
* Tumor progression after receiving standard/approved chemotherapy or where there is no approved therapy.
* One or more tumors measurable on radiograph or CT scan, or evaluable disease (e.g., malignant ascites).
* Karnofsky performance status of greater than or equal to 70.
* Life expectancy of at least 3 months.
* Age at least 18 years.
* Patients must have central IV access, or agree to the insertion of a central IV line.
* Normal oxygen saturation by pulse oximetry on room air
* A negative pregnancy test (if female).
* Acceptable liver function as evaluated by laboratory results
* Acceptable renal function as evaluated by laboratory results
* Acceptable hematologic status as evaluated by laboratory results
* No clinically significant urinalysis abnormalities
* Acceptable coagulation status as evaluated by laboratory results
* Fertile men and women must use effective contraceptive methods during the study.

Exclusion Criteria:

* Seizure disorders requiring anticonvulsant therapy.
* Known brain metastases (unless previously treated and well controlled for a period of greater than or equal to 3 months).
* Severe chronic obstructive pulmonary disease with hypoxemia, or an uncorrectable pulmonary compromise.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to the first dose of test drug.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Pregnant or nursing women.
* Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within one month prior to study entry (6 weeks for nitrosoureas or Mitomycin C).
* Unwillingness or inability to comply with procedures required in this protocol.
* Known infection with HIV, hepatitis B, or hepatitis C.
* Clinically significant bleeding event within the last 3 months, unrelated to trauma, or underlying condition that would be expected to result in a bleeding diathesis.
* Patients who are currently receiving any other investigational agent.
* Patients who have exhibited allergic reactions to a similar structural compound (e.g., fluoroquinolones, biological agent or formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and Dose limiting toxicity (DLT) | Cycle 1
Recommended Phase 2 dose | Cycle 1

SECONDARY OUTCOMES:
Pharmacokinetics (PK) in humans of intravenously administered quarfloxin | One month
Evaluation of antitumor activity of quarfloxin by objective radiologic assessment | Every 2 months
Pharmacodynamic evaluation of antitumor activity | Monthly

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Scottsdale, Arizona
  - San Antonio, Texas